CLINICAL TRIAL: NCT05287542
Title: Releasing Residual Cognitive Capacity After Acquired Brain Injury: A Randomized Controlled Trial Using Hypnotic Suggestion in Rehabilitation of Working Memory
Brief Title: Hypnosis in Working Memory Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnaas Rehabilitation Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hypnoseprosjektet
Record Dates: First submitted 2022-03-09; First posted 2022-03-18 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Cognitive Rehabilitation; Brain Injuries; Cognitive Impairment; Working Memory
Keywords: Aquired brain injury; Rehabilitation; Randomized controlled trial (RCT); Clinical Hypnosis; Self-efficacy
MeSH Terms: conditions — Brain Injuries; Cognitive Dysfunction | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: It is not possible to blind participants or therapists to group allocation during the intervention. Independent Outcome Assessor(s) will be blinded to group allocation. Participants will be provided with new IDs in final database, blinding researchers to which group is the interventions group, active control group or passive control group during analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hypnotic suggestion (Experimental): During the first phase of the study, two groups will receive identical hypnotic inductions followed by targeted suggestion for one group and non-targeted suggestion for the other. The targeted procedure consists of suggestions about enhancing WM functions through the instantiation of preinjury WM ability in the present using age regression and visualizations of brain plasticity.
  Interventions: Other: Hypnotic suggestion
- Mindfulness (Active Comparator): The targeted procedure consists of suggestions about enhancing WM functions through the instantiation of preinjury WM ability in the present using age regression and visualizations of brain plasticity.
  Interventions: Other: Mindfulness
- No treatment (No Intervention): The passive control group receives no intervention

INTERVENTIONS:
Other: Hypnotic suggestion — The intervention group will receive four weekly 60 min. sessions with hypnosis treatment including induction followed by hypnotic suggestion.
  Arms: Hypnotic suggestion
Other: Mindfulness — The active control group will receive four weekly 60 min. sessions of induction and mindfulness-based instructions.
  Arms: Mindfulness

SUMMARY:
Establishment of effective, efficient, and evidence-based interventions in rehabilitation of working memory (WM) deficits after acquired brain injury (ABI) is sorely needed. Despite robust evidence for the usefulness of clinical hypnosis in a wide range of clinical conditions, and improved understanding of mechanisms underlying it ́s effects, the potential of clinical hypnosis in cognitive rehabilitation is virtually unexplored. The current study seeks to replicate resent intriguing findings where large effects of hypnotic suggestion were seen on WM capacity following ABI, and further, explore underlying mechanisms of change.

DETAILED DESCRIPTION:
The potential impact of applying hypnosis in cognitive rehabilitation is substantial. Deficits in WM is one of the most common challenges after ABI and plays a critical role in post-injury outcome. Still, state-of-the-art approaches within WM rehabilitation have not been able to produce significant effects that transfer to real- life functioning for the affected patients. Building on the strong results of hypnosis on WM in ABI from a Danish single trial, we will aim at replication and expansion of the study in a Norwegian context. The initial study will be expanded in terms of number of participants, injury-characteristics will be included, outcome measures of relevance to real-life functioning, and underlying mechanisms of change will be explored. Self-efficacy is generalizable by nature (self-efficacy gained from mastery experiences in one situation generalizes to others), thus WM rehabilitation effects are expected to generalize and transfer to other domains in daily life.

This randomized controlled trial (RCT) aims to evaluate the effectiveness of hypnosis in WM rehabilitation in ABI patients. Ninety patients will be recruited from Sunnaas Rehabilitation Hospital. Inclusion criteria are non-progressive ABI, minimum 12 months post- injury, ongoing WM deficits and age between 18 and 67 years. Patients will be randomized to either a) an intervention group receiving four weekly 60 min. sessions with induction and hypnosis, b) an active control group receiving four weekly 60 min. sessions of induction and mindfulness, or c) a passive control group without intervention. The targeted procedure consists of suggestions about enhancing WM functions through the instantiation of preinjury WM ability in the present using age regression and visualizations of brain plasticity. The non- targeted suggestions contain no explicit mentioning of ABI or WM-related abilities. Each participant will be assessed at baseline, immediately after intervention and six months after baseline. Primary outcome is WM as measured by neuropsychological tests as well as self- and informant reported WM capacity. Secondary outcomes include self-rated ABI related symptoms, self-efficacy, mental health, and global outcome. A process evaluation will be carried out to evaluate treatment experience,

Rehabilitation of impaired WM after ABI has hitherto yielded limited clinical effects, and clinical trials of new interventions are thus warranted. Long-standing empirical evidence demonstrates that hypnosis is an effective therapeutic technique in a wide range of conditions, including in altering cognitive functions and improving WM in healthy adults, supported by imaging data. Recent exploratory research has suggested remarkable efficacy of hypnosis in improving WM in patients with ABI. However, these findings need replication in studies applying scientifically rigorous designs. If successful, our ambition is to provide recommendations and materials to implement hypnotic suggestion as an adjunct treatment following ABI in Norwegian rehabilitation clinics. Study findings may inform future studies exploring the use of clinical hypnosis in other areas of rehabilitation, such as mild TBI, and in other neurological conditions where WM deficit is prominent.

ELIGIBILITY:
Inclusion Criteria:

* A documented non-progressive ABI, minimum 12 months post- injury and ongoing WM deficits by self-report and/or neuropsychological assessment
* The above mentioned patients have received multidisciplinary cognitive rehabilitation before participation

Exclusion Criteria:

* Patients with severe mental illness
* Patients progressive neurologic disease
* Patients with ongoing ICD-10 diagnosis of substance dependence
* Patients that lack Norwegian language skills

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in WM on neuropsychological tests | Change from Baseline (T1) to immediately after the intervention period (T2) and 8 months after Baseline (T3)
  Measured by the WM Index WAIS IV
Change in WM-related symptoms in everyday life | Change from Baseline (T1) to immediately after the intervention period (T2) and 8 months after Baseline (T3)
  Assessed with the WM subscale from the Behavior Rating Inventory of Executive functioning Adult version (BRIEF-A) on a 3-point scale: Never a problem, sometimes a problem or often a problem. Higher scaled score indicates higher level of problems with WM.

SECONDARY OUTCOMES:
Change in cognitive composite score as seen on neuropsychological tests | Change from Baseline (T1) to immediately after the intervention period (T2) and 8 months after Baseline (T3)
  Measured by Trail Making A+B, D-KEFS CWIT 1-4, CVLT-II, WAIS IV Digit Symbol
Change in TBI related challenges in everyday life | Change from Baseline (T1) to immediately after the intervention period (T2) and 8 months after Baseline (T3)
  Measured by the Patient Competency Rating Scale on a 5-point scale from 1 can't do it to 5: No problem to do it. Higher total scaled score represents better every day functioning.
Change in self reported mental health | Change from Baseline (T1) to immediately after the intervention period (T2) and 8 months after Baseline (T3)
  Measured with the Hopkins Symptom Checklist (HSCL) on a scale from 1 (not at all) to 4 (a lot). Higher mean score reflects a higher level of emotional distress.
Change in quality of life | Change from Baseline (T1) to immediately after the intervention period (T2) and 8 months after Baseline (T3)
  Assessed with Quality of Life After Brain Injury (QOLIBRI) on a satisfaction scale from 0 (not satisfied) to 5 (very satisfied). Higher satisfaction indicates higher quality of life.
Changes in community integration | Change from Baseline (T1) to immediately after the intervention period (T2) and 8 months after Baseline (T3)
  Assesed with Participation Assessment with Recombines Tools-Objective (PART-O) on a 5-point scale: None, 1-4 hours, 5-9 hours, 10-19 hours, 20-34 hours, 35 hours or more. Higher mean scaled score indicates better community integration.

OTHER OUTCOMES:
Changes in ABI related self-efficacy | Change from Baseline (T1) to immediately after the intervention period (T2) and 8 months after Baseline (T3)
  The tool to measure Traumatic Brain Injury Self-Efficacy is rated on a scale from 0 (very uncertain) to 10 (Very certain). Higher total score on the questionnaire indicates higher TBI related self-efficacy.
Changes in WM self-efficacy | Change from Baseline (T1) to immediately after the intervention period (T2) and 8 months after Baseline (T3)
  The Memory Self-Efficacy Questionnaire (MSEQ) is rated on a scale from 0 (never) to 12 (100% of the time). Higher total scales score indicates higher WM self-efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Løvstad, Profesor, Principal Investigator — Sunnaas Rehabilitation Hospital and University of Oslo
Locations (1):
- Sunnaas Rehabilitation Hospital, Nesoddtangen, Akershus, Norway

REFERENCES:
- [Derived] Eide LS, Rike PO, Reme SE, Snekkevik H, Rossner S, Rosen G, Lindelov JK, Lovstad M. Using hypnotic suggestion in the rehabilitation of working memory capacity after acquired brain injury: study protocol for a randomized controlled trial. Trials. 2024 Jan 2;25(1):11. doi: 10.1186/s13063-023-07867-z. PMID 38167204